CLINICAL TRIAL: NCT06093711
Title: The Prevalence, Type, And Risk Factors of Urinary Incontinence in Married Women and Its Effect on Their Quality of Life
Brief Title: Urinary Incontinence in Married Women
Status: Completed | Type: Observational
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, MAHİNUR DURMUŞ İSKENDER, Assistant Professor, Kastamonu University
Other Study IDs: MDURMUSISKENDER
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Description — All patients were briefed about the research purpose and procedure. They were also informed about the following points: (1) participation is voluntary, (2) they can withdraw from the study at any stage without explanation, (3) the data will be used only for scientific purposes and will not be shared with third parties, and (4) they will remain anonymous throughout the research. Informed consent was obtained from those who agreed to participate. It took each participant 20-25 minutes to fill out the data collection tools.

SUMMARY:
Background: Urinary incontinence is involuntary urinary leakage. Although it is not life-threatening, it dramatically influences the quality of life. This study was conducted to determine the prevalence, type, and risk factors of UI in married women and its effect on their quality of life.

Methods: This descriptive and cross-sectional study was conducted on 413 women. This research was conducted between October 2022 and July 2023 in the central district of a province in the northwestern region of Türkiye. The data were collected using a Personal Information Form and the Incontinence Quality of Life. The data were analyzed using the Statistical Package for Social Sciences (SPSS for Windows, IBM, version 22.0) at a significance level of 0.05. Descriptive statistics baseline characteristics. Normality was tested using the Kolmogorov-Smirnov test. The results showed that the data were normally distributed. Therefore, an independent t-test (t-table value) was used for two independent groups, while an Analysis of Variance (ANOVA) (F-table value) was used for more than two groups.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is involuntary urinary leakage. This condition causes physical, psycho-social, and economic problems.1 It is more prevalent in women than in men. It occurs in women during pregnancy, childbirth, or menopause. It can also be triggered by factors such as advanced age, diabetes mellitus, chronic urinary infections, hysterectomy, and obesity.2,3 While urinary incontinence is not a life-threatening condition, it significantly impacts the quality of life for women. It leads to social phobia, social isolation, reduced self-confidence and self-esteem, embarrassment, psychological issues, as well as individual and societal costs.2-4 Urinary incontinence represents a growing burden in numerous countries.5 (Milsom et al., 2014).

Urinary incontinence constitutes a significant public health issue when considering the global female population, their participation in the workforce, and their role in social life.6 Urinary incontinence afflicts more than 40% of women worldwide.7 (Liu et al., 2014). The prevalence of UI is 48.3%, 46.4%, 31.9%, and 18.7% in women over 18 years of age living in Germany, Denmark, China, and Norway, respectively.8-10 The prevalence of UI is 23.6% in women aged 45-60 years living in Brazil.11 The prevalence of UI ranges from 16.4% and 49.7 in Turkish women.12 The projected number of women with UI in the United States is expected to reach 28.4 million by 2050.13 Investigators believe that the prevalence of UI may be underestimated because many women either seek healthcare assistance late or not at all due to perceiving it as a natural consequence of aging or childbirth or because they feel embarrassed about the issue. Furthermore, only a small fraction of women who are diagnosed with UI receive effective treatment.2,3,14 More than half of women with UI (66.4%) take approximately three years to seek medical assistance due to fears of stigmatization and a lack of information about treatment.4,15 The treatment and care for UI necessitate a multidisciplinary approach due to the complexity of the condition and the various issues it involves. However, before women are willing to seek medical assistance for UI, they must first recognize it as a medical issue. Hence, it is essential to develop a comprehensive understanding of UI, raise awareness among women about the condition, and provide ongoing support for those affected by it. By taking these steps, we can effectively manage and prevent this condition, as well as create opportunities for early diagnosis and treatment. Therefore, this study investigated the prevalence, type, and risk factors of UI in married women and its effect on their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years, married women, Those who agreed to participate in the research.

Exclusion Criteria:

* she wants to leave the research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Married women will be included.
Study Population: The study population consisted of all married women in the central district of a province in the northwestern region of Türkiye. The sample size was calculated using the formula for a known population. The results showed that a sample of 382 would be large enough to detect significant differences. The sample consisted of 413 women who agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Incontinence Quality of Life | October 2022 and July 2023
  Incontinence Quality of Life The total score ranges from 22 to 110, with higher scores indicating a higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No